CLINICAL TRIAL: NCT03971279
Title: Long Term Efficacy of Dexamethasone Intravitreal Implant (Ozurdex®) in Treatment of Recurrent VKH Uveitis
Brief Title: Dexamethasone Intravitreal Implant (Ozurdex®) for Recurrent Vogt-Koyanagi-Harada (VKH) Disease Posterior Uveitis
Status: Completed | Type: Observational
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Tarek Roshdy mohamed Mahgoub ELhamaky, Lecturer of ophthalmology, Benha University
Other Study IDs: hamaky2
Record Dates: First submitted 2019-05-30; First posted 2019-06-03 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Posterior Uveitis
Keywords: dexamethasone;VKH
MeSH Terms: conditions — Uveitis, Posterior | interventions — Calcium Dobesilate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Dexamethasone Ophthalmic implant — intravitreal injection of ozurdex implant
  Other Names: ozurdex implant

SUMMARY:
VKH disease is a vision threatening condition.The investigators consider that ozurdex intravitreal implant is an effective line of treatment in recurrent VKH posterior uveitis.

DETAILED DESCRIPTION:
Baseline ,and postoperative 1 ,6 ,12 and 24 months full ophthalmic examination was done.

Procedure included intravitreal injection of Dexamethasone implant 0.7 mg (Ozurdex(®); Allergan, Inc, Irvine, CA)

ELIGIBILITY:
Inclusion Criteria:

* Recurrent VKH posterior uveitis

Exclusion Criteria:

* retinal pathology, other causes of posterior uveitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 16 patient with VKH disease who have recurrent attacks of posterio uveitis
Sampling Method: Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-11-22 (Actual); Study Completion 2019-11-22 (Actual)

PRIMARY OUTCOMES:
Best corrected visual acuity (BCVA) | 2 years
  Change in BCVA

SECONDARY OUTCOMES:
optical coherence tomography (OCT) foveal thickness | 2 years
  changes in central foveal thickness

CONTACTS AND LOCATIONS:
Overall Officials: Tarek Elhamaky, Principal Investigator — Benha university faculty of medicine , INMC
Locations (1):
- INMC, Abu Dhabi, United Arab Emirates